CLINICAL TRIAL: NCT01816659
Title: An Open-Labeled Pilot Study of Biomarker Response in Patients With Colorectal Cancer or Endoscopically Non-Resectable Adenomas Following Short-Term Exposure to Metformin Extended Release (ER)
Brief Title: An Open-Labeled Pilot Study of Biomarker Response Following Short-Term Exposure to Metformin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2012-1150; NCI-2013-00994 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Carcinoma
Keywords: Colorectal Carcinoma; Endoscopically Non- Resectable Adenomas; Colonic lesion; Biomarker; Metformin-ER; Metformin; Extended release; Colonoscopy; Colon cancer surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin + Colon Surgery (Experimental): Patients randomized to Metformin-ER 500 mg once daily for one week and then escalation to 1000 mg/day for the duration of the trial. The duration of the trial will be from the preoperative endoscopy till the surgery, and should be not less than 10 days and not more than 30 days.
  Interventions: Drug: Metformin ER
- Colon Surgery Alone (No Intervention): Patients will not receive any study drug from the time of colonoscopy until surgery.

INTERVENTIONS:
Drug: Metformin ER — 500 mg by mouth once daily, beginning the day after colonoscopy for one week, and then escalation to 1000 mg/day. The duration of the trial will be from the preoperative endoscopy till the surgery, and should be not less than 10 days and not more than 30 days.
  Other Names: Metformin
  Arms: Metformin + Colon Surgery

SUMMARY:
The goal of this clinical research study is to learn more about the possible effects of metformin extended release (ER) in patients with colon cancer or adenomas who are about to have surgery. The safety of this drug will also be studied.

Metformin-ER is commonly used to control blood sugar levels in patients with diabetes. It is also designed to block a protein in tumor cells that is important in tumor growth and blood vessel development. This may cause cell death or reduce the spread of the disease.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

* If you are in Group 1, you will receive metformin ER. You will have a 2 in 3 chance of being assigned to Group 1.
* If you are in Group 2, you will receive no treatment. You will have a 1 in 3 chance of being assigned to Group 2.

Study Drug Administration:

If you are in Group 1, You will start taking the drug the day after your colonoscopy (or later if your surgery is scheduled to be more than 30 days after the colonoscopy) and will continue to take it until your scheduled surgery (for up to 30 days). During the first week you will take one tablet of metformin-ER by mouth one time each day with food. From the beginning of the second week until your scheduled surgery, you will take two tablets of metformin-ER by mouth one time each day with food. If you have side effects, your dose may be lowered.

If you are in Group 2, you will not receive any study drug from the time of your colonoscopy until surgery.

Study Visits:

On the day of your colonoscopy:

* Your medical history will be recorded and you will be asked about any drugs you may be taking.
* You will have a physical exam.
* Extra tissue samples will be collected during the colonoscopy for routine and biomarker testing. Biomarkers are small pieces of material or substances found in you tissue that may provide information about your condition or the disease.
* The study staff will call you 1 week after your colonoscopy and ask about your general health and about any side effects you may be having.

On the day before surgery or the day of the surgery itself:

* Your weight will be measured.
* Blood (about 3 tablespoons) will be drawn for routine tests and for research about the safety of metformin-ER and how it may affect the disease. This routine blood draw will include a pregnancy test if you are able to become pregnant.
* You will be asked about your general health and about any side effects you may be having.
* During the surgery, extra tissue samples will be collected for biomarker testing.

Length of Study:

You will be on study for up to 30 days. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have had the surgery.

This is an investigational study. Metformin-ER is FDA approved and commercially available for the treatment of type 2 diabetes. Its use in this study is investigational.

Up to 23 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18- 75 years
2. Colonic lesion that should be removed surgically:
3. 2.a. CRC that is potentially resectable and not requiring neoadjuvant treatment.
4. 2.b. Endoscopically non-resectable adenoma.
5. 2.c. Familial Adenomatous Polyposis (FAP) patient that requires colectomy or proctocolectomy.
6. Need for perioperative colonoscopy as a part of standard of care evaluation:
7. 6.a. CRC or adenoma for which the colorectal surgeon requires a preoperative colonoscopy or sigmoidoscopy for any reason, including but not limited to:
8. 6.a.a. No outside colonoscopy
9. 6.a.b. No outside pathology
10. 6.a.c. Partially obstructing tumor or
11. 6.a.d. Otherwise unsatisfactory outside colonoscopy
12. 6.a.e. Rectal cancer requiring EUS
13. 6.a.f. Second opinion on adenoma regarded as endoscopically non-resectable on outside colonoscopy; or
14. 6.b. Patient found on initial MDACC colonoscopy to have CRC or endoscopically non-resectable adenoma, most commonly patients undergoing average or high risk (familial, history of adenoma) screening colonoscopy.
15. Ability to give informed consent.
16. Diabetic patients are eligible but they may be excluded if they are taking Metformin, insulin or sulfonylureas.

Exclusion Criteria:

1. Patients with renal insufficiency defined as serum creatinine >= 1.4 mg/dl for females and >= 1.5 mg/dl for males
2. Pregnant or nursing women
3. A malignancy currently under active therapy
4. Unstable angina
5. Uncontrolled ischemic cardiac disease or symptomatic congestive heart failure (e.g. Class III or IV New York Heart Association's Functional Classification)
6. Current usage of Metformin
7. Current usage of insulin, sulfonylureas
8. History of lactic acidosis
9. Chronic liver disease or cirrhosis
10. Inability to give informed consent
11. Other investigational drugs within the past one year or concurrently
12. Known hypersensitivity or intolerance to Metformin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Comparison of Ki-67 in Tumor Samples | 2 weeks
  Primary outcome measure is change in the percentage of Ki67-positive-staining cells between the baseline colonoscopy and surgery in the colon rectal cancer/non-resectable adenoma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lynch, MD, JD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org